CLINICAL TRIAL: NCT00831506
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Two-Way Crossover Study To Evaluate The Steady-State Effect Of Dimebon (PF-01913539) On The Safety, Tolerability, And Steady-State Pharmacokinetics Of Digoxin In Healthy Subjects
Brief Title: Dimebon (PF-01913539)-Digoxin Drug-Drug Interaction Study In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B1451021
Record Dates: First submitted 2009-01-27; First posted 2009-01-29 (Estimated); Last update posted 2009-06-12 (Estimated); Status verified 2009-06

CONDITIONS: Alzheimer Disease; Huntington Disease
Keywords: digoxin dimebon drug-drug interaction study
MeSH Terms: conditions — Alzheimer Disease; Huntington Disease | interventions — Digoxin; latrepirdine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): digoxin once daily (0.125 mg QD) plus placebo three times daily (TID), 8 hours apart for 14 days.
  Interventions: Drug: digoxin
- B (Experimental): digoxin once daily (0.125 mg QD) plus Dimebon three times a day, 8 hours apart for 14 days (10 mg TID on Days 1-7 and 20 mg TID on Days 8-14).
  Interventions: Drug: digoxin; Drug: dimebon

INTERVENTIONS:
Drug: digoxin — digoxin once daily (0.125 mg QD) plus placebo three times daily (TID), 8 hours apart for 14 days.
  Arms: A
Drug: digoxin — digoxin once daily (0.125 mg QD) for 14 days.
  Arms: B
Drug: dimebon — Dimebon three times a day, 8 hours apart for 14 days (10 mg TID on Days 1-7 and 20 mg TID on Days 8-14).
  Arms: B

SUMMARY:
This study has been designed to confirm, in healthy subjects, the lack of a clinically important pharmacokinetic interaction between Dimebon, at the proposed maximum commercial dose of 20 mg TID (administered every 8 hours), and digoxin (Lanoxin®) 0.125 mg QD, a sensitive P-gp substrate recommended by FDA.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* A known history of hypersensitivity or previous intolerance to Dimebon or digoxin.
* Evidence or history of clinically significant hematological, renal, endocrine,pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic,seasonal allergies at time of dosing) disease or clinical findings at screening.
* Pregnant or nursing women; women of childbearing potential (WOCBP) who are unwilling or unable to use an acceptable method of contraception as outlined in the protocol from at least 14 days prior to the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
AUC24 and Cmin of digoxin on Day 14 | Day 14

SECONDARY OUTCOMES:
Cmax, Tmax, Ae, and renal clearance of digoxin on Day 14 | Day 14
Adverse event monitoring through Day 14 including physical/neurological examination findings | Day 14
Clinical safety assessments through Day 14 including chemistry, hematology, and vital signs | Day 14
12-lead ECGs through Day 14 | Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1451021&StudyName=Dimebon%20%28PF-01913539%29-Digoxin%20Drug-Drug%20Interaction%20Study%20In%20Healthy%20Subjects